CLINICAL TRIAL: NCT01622465
Title: Effect of Cycle Ergometer in the Rehabilitation of Elderly Patients With Total Hip Arthroplasty: Randomized Controlled Trial
Brief Title: Effect of Cycle Ergometer in the Rehabilitation of Elderly Patients With Total Hip Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Mariana Katia Rampazo, Principal Investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 403/2011
Record Dates: First submitted 2012-06-11; First posted 2012-06-19 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Osteoarthritis, Hip; Osteonecrosis
Keywords: Hip arthroplasty; Aged; Rehabilitation; Exercise therapy
MeSH Terms: conditions — Osteoarthritis, Hip; Osteonecrosis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ergometer cycling (Experimental): Patients will participate of the exercises program with ergometer cycling and conventional exercises.
  Interventions: Behavioral: Ergometer cycling
- Conventional exercises (Active Comparator): Patients will participate only of the conventional exercises program.
  Interventions: Behavioral: Conventional exercises

INTERVENTIONS:
Behavioral: Ergometer cycling — Patients will participate of the exercises program with ergometer cycling and conventional exercises. The program will initiate after two weeks of the postoperative and will continue until three months of the postoperative
  Arms: Ergometer cycling
Behavioral: Conventional exercises — Patients will participate only of the conventional exercises program. The program will initiate after two weeks of the postoperative and will continue until three months of the postoperative
  Arms: Conventional exercises

SUMMARY:
The aim of this study is to evaluate the effects of an exercise program with a cycle ergometer in functional outcome and related-health quality of life (RHQL) in elderly patients with total hip arthroplasty.

DETAILED DESCRIPTION:
Behavioral: Ergometer Cycling Ergometer Cycling under the guidance of a physical therapist after the second postoperative week. These training sessions were scheduled to be performed two times a week for a time period of at least eith weeks.

Behavioral: No ergometer cycling Patients of the no ergometer cycling group did not receive any ergometer cycling after surgery, only conventional exercises.

ELIGIBILITY:
Inclusion Criteria:

* Aged patients (60 years or more) of both sexes
* Being submitted to the total hip arthroplasty, primary and unilateral, for hip osteoarthritis or hip osteonecrosis
* no history of physical therapy two months before surgery

Exclusion Criteria:

* arthroplasty of hip fracture or other condition;
* neurological disease that compromises motor function;
* postoperative complications (dislocation, infection, cardiovascular events);
* revision of the prosthesis;
* patients who are unable to attend the sessions of physical therapy or refused to participate in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hip function at three months | Baseline and three months
  Harris Hip Score (HHS) will be used to collect the data at baseline and at three months

SECONDARY OUTCOMES:
Change from baseline in physical performance of lower limbs at three months. | Baseline and three months
  "Short Physical Performance Battery (SPPB)" developed by Guralnik (1994), to evaluate of balance, gait speed and muscle strenght, of lower limbs will be used to collect the data at baseline and at three months.
Change from baseline in health-related quality of life (HRQOL)at three months by generic questionnaire | Baseline and three months
  The generic questionnaire evaluation HRQOL "Medical Outcomes Survey 36 - Item Short-Form" developed by Ware and Sherboune (1992) will be used to collect the data at baseline and at three months
Change from baseline in health-related quality of life (HRQOL) at three months by specific questionnaire | Baseline and three months
  The specific questionnaire evaluattion HRQOL "Western Ontario and McMaster Universities (WOMAC)" developed by Bellamy (1988) will be used to collect the data at baseline and at three months.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana K Rampazo, PhDCandidate, Principal Investigator — University of Campinas, Nursing Department; Maria José D'Elboux, PhD, Study Chair — University of Campinas, Nursing Department
Locations (1):
- Hospital das Clínicas da Universidade Estadual de Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Rampazo-Lacativa MK, D'Elboux MJ. Effect of cycle ergometer and conventional exercises on rehabilitation of older patients with total hip arthroplasty: study protocol for randomized controlled trial. Trials. 2015 Apr 8;16:139. doi: 10.1186/s13063-015-0647-8. PMID 25873151